CLINICAL TRIAL: NCT05105451
Title: Study on the Characteristics of Non-targeted Metabolomics and EEG of Delayed Neurocognitive Recovery in Elderly Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Other Study IDs: SH9H-2021-T120
Record Dates: First submitted 2021-05-28; First posted 2021-11-03 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Delayed Neurocognitive Recovery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients in the control group were followed up without dNCR postoperatively.: If the MOCA or MMSE assessment all show a negative resluts at all time point.
  Interventions: Other: Collecting clinical data, EGG，arterial blood gas data and venous blood sample
- Patients in the case group were followed up with dNCR postoperatively.: If the MOCA assessment is positive at any time point after surgery, and there is a positive MMSE at any time point after surgery(no need for both MOCA and MMSE to be positive at the same time), it is defined as the occurrence of dNCR.
  Interventions: Other: Collecting clinical data, EGG，arterial blood gas data and venous blood sample

INTERVENTIONS:
Other: Collecting clinical data, EGG，arterial blood gas data and venous blood sample — Collecting clinical data(before induction of anesthesia and first day after surgery), EGG（first day after surgery），arterial blood gas data(before induction of anesthesia and first day after surgery) and venous blood sample （before induction of anesthesia and first day, third day and 7th day after surgery）

SUMMARY:
Perioperative neurocognitive disorder (PND) refers to a broad range of postoperative cognitive complications, including preoperatively diagnosed cognitive decline, postoperative delirium (POD), delayed neurocognitive recovery (dNCR), and neurocognitive disorders . Among them, dNCR refers to a decline in cognitive function that occurs approximately 1-4 weeks after anesthesia/surgery in elderly patients. It is associated with an increased risk of postoperative complications and an increased length of hospital stay.

The identification of potential predictive biomarkers would be beneficial for determining the individual risk of developing dNCR and for postoperative management of elderly patients. Although some predictive markers for PNDs, such as inflammatory factors, tau protein, S100B protein, neuron-specific enolase, and brain-derived neurotrophic factor, are widely known, most of them are postoperative predictive markers. The markers that can be used to predict PNDs before anesthesia/surgery are still largely unknown.

Preoperative markers allow us to identify individuals who are susceptible to dNCR and intervene early. It is unclear whether the metabolic status of preoperative patients is related to the occurrence of postoperative cognitive dysfunction (POCD). In the framework of systems biology based on genome, transcriptome, proteome, and metabolome, metabolomics is the closest to biological phenotypes because it reflects biological events that have occurred in living organisms. Considering that metabolome reflects the metabolites of all biochemical reactions that have already taken place in an organism and contains a huge amount of information about an organism's health, preoperative patient metabolites may be a useful predictive biomarker. In this study, we used serum metabolomics to develop non-invasive, easily detectable, and inexpensive preoperative biomarkers from patient blood to determine the individual risk of dNCR and the relationship between metabolic system abnormalities and the pathogenesis of dNCR.

ELIGIBILITY:
Inclusion Criteria:

* Gender: no gender limit
* 65 years or older .
* Complete the operation in our hospital
* ASA classification I-II level
* Agree to participate in this research and agree to sign an informed consent form

Exclusion Criteria:

* History of preoperative psychosis and psychotropic drug use
* The subject is diagnosed with AD;
* Abnormal preoperative mental scale assessment
* Have a history of emergency rescue during the perioperative period

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Our research is a single center, nested case-control study. Preoperatively collect the information of the elderly patients over 65 years old without undergoing craniocerebral operations, including the vital signs, the examination reports and other related data after excluding the factors that can't be included in the group. The patients' health scales and dNCR. scales were evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-05-22 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
MMSE (mini-mental state examiniation) | 1 day after surgery
  MMSE scale score, If the MMSE assessment is positive at any time point, and there is a positive MMSE at any time point (no need for both MOCA and MMSE to be positive at the same time), it is defined as the occurrence of dNCR.
MOCA (Montreal Cognitive Assessment) | 1 day after surgery
  MOCA sacle score, If the MOCA assessment is positive at any time point, and there is a positive MMSE at any time point (no need for both MOCA and MMSE to be positive at the same time), it is defined as the occurrence of dNCR.
MMSE (mini-mental state examiniation) | 3 day after surgery
  MMSE scale score, If the MMSE assessment is positive at any time point, and there is a positive MMSE at any time point (no need for both MOCA and MMSE to be positive at the same time), it is defined as the occurrence of dNCR.a positive MMSE at any time point (no need for both MOCA and MMSE to be positive at the same time), it is defined as the occurrence of dNCR.
MOCA (Montreal Cognitive Assessment) | 3 day after surgery
  MOCA sacle score, If the MOCA assessment is positive at any time point, and there is a positive MMSE at any time point (no need for both MOCA and MMSE to be positive at the same time), it is defined as the occurrence of dNCR.
MMSE (mini-mental state examiniation) | 7 day after surgery
  MMSE scale score, If the MMSE assessment is positive at any time point, and there is a positive MMSE at any time point (no need for both MOCA and MMSE to be positive at the same time), it is defined as the occurrence of dNCR. a positive MMSE at any time point (no need for both MOCA and MMSE to be positive at the same time), it is defined as the occurrence of dNCR.
MOCA (Montreal Cognitive Assessment) | 7 day after surgery
  MOCA sacle score, If the MOCA assessment is positive at any time point, and there is a positive MMSE at any time point (no need for both MOCA and MMSE to be positive at the same time), it is defined as the occurrence of dNCR.
MOCA (Montreal Cognitive Assessment) | right before surgery
  MOCA sacle score,baseline
MMSE (mini-mental state examiniation) | right before surgery
  MMSE scale score, baseline
T-MoCA (The telephone MoCA) | 15 day after surgery
  MOCA sacle score, If the MOCA assessment is positive at any time point, and there is a positive MMSE at any time point (no need for both MOCA and MMSE to be positive at the same time), it is defined as the occurrence of dNCR.
T-MoCA (The telephone MoCA) | 30 day after surgery
  MOCA sacle score, If the MOCA assessment is positive at any time point, and there is a positive MMSE at any time point (no need for both MOCA and MMSE to be positive at the same time), it is defined as the occurrence of dNCR.

SECONDARY OUTCOMES:
3D-CAM | 1 day after surgery
  3D-CAM score
Self-Rating Anxiety Scale | right before surgery
  Self-Rating Anxiety Scale score
Self-rating depression scale | right before surgery
  Self-rating depression scale score

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jiang, Doctor, Study Director — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai 9Th Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang L, Liu J, Zhou R, Liu J, Zhang J, Mao H, Yan J, Jiang H. Preoperative tyrosine is associated with postoperative delayed neurocognitive recovery in elderly: Evidence from two hospitals. Clin Nutr ESPEN. 2025 Aug;68:727-736. doi: 10.1016/j.clnesp.2025.06.016. Epub 2025 Jun 13. PMID 40518008
- [Derived] Mao H, Huang H, Zhou R, Zhu J, Yan J, Jiang H, Zhang L. High preoperative blood oxaloacetate and 2-aminoadipic acid levels are associated with postoperative delayed neurocognitive recovery. Front Endocrinol (Lausanne). 2023 Jul 31;14:1212815. doi: 10.3389/fendo.2023.1212815. eCollection 2023. PMID 37583434

DOCUMENTS (1):
  • Informed Consent Form (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT05105451/ICF_000.pdf